CLINICAL TRIAL: NCT03998527
Title: Non-Invasive Spinal Cord Stimulation and Respiratory Plasticity
Brief Title: Non-Invasive Spinal Cord Stimulation After Injury
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Alexander V Ovechkin, MD, PhD, Assoc Professor, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 17.1279
Record Dates: First submitted 2019-06-20; First posted 2019-06-26 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Spinal Cord Injuries
Keywords: Respiration; Motor control
MeSH Terms: conditions — Spinal Cord Injuries; Respiratory Aspiration

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Non-Disabled (ND) and Spinal Cord Injured (SCI) controls (Experimental): The ND Control group (n=6) and SCI Control group (n=6) will be used to assess related values as acute effects of transcutaneous electrical spinal cord stimulation (TcESCS) itself and will not receive any training intervention. The ND group will receive baseline assessments, then up to 12 (4-Respiratory function, 4-Arm function, and 4-Trunk function) TcESCS mapping experiments, followed by repeating the assessments in the presence of TcESCS. The investigators will decide which stimulation type should be used for the post-mapping assessments.
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation (TcESCS)
- Spinal Cord Injured (SCI) intervention groups (Experimental): The respiratory training (RT) group (n=6) will receive the respiratory training intervention only); the transcutaneous electrical spinal cord stimulation (TcESCS) group (n=6) will receive transcutaneous spinal cord stimulation only; TcESCS + RT group (n=6) will receive TcESCS combined with RT; TcESCS + Arm Training (AT) group (n=6) will receive TcESCS combined with AT; and TcESCS + Trunk Training (TT) group (n=6) will receive TcESCS combined with TT.
  Interventions: Device: Transcutaneous Electrical Spinal Cord Stimulation (TcESCS)

INTERVENTIONS:
Device: Transcutaneous Electrical Spinal Cord Stimulation (TcESCS) — TcESCS is a non-invasive DC battery powered device. Investigators and/or research team members will continually assess the appropriate stimulation parameters including configurations, current, voltage and frequency delivered by up to five active electrodes applied on skin of the back from cervical to lumbar levels. Stimulation parameters used during experimental assessments and interventions will be closely monitored by the research team. Every research participant will be slowly acclimated to stimulation. Blood pressure, heart rate, respiratory rate, and electromyography will be closely monitored while we are determining the correct stimulation parameters in the lab. During the stimulation training sessions, we will monitor blood pressure regularly throughout the session.
  Other Names: Non-invasive spinal cord stimulation

SUMMARY:
The goal of this study is to assess the function of the lungs and the muscles are used to breathe after individuals receive respiratory training, spinal cord stimulation, a combination of respiratory training and stimulation, a combination of arm training and stimulation, or a combination of trunk training and stimulation. The respiratory, arm, and trunk training combined with the spinal stimulation interventions are being used to activate the spinal cord below the level of injury. Investigators will be looking for changes in the function of the lungs and trunk muscles before, during, and after these task-specific and non-task-specific interventions for breathing to determine which one has the greatest effect. The results of this study may aid in the development of treatments to help individuals with spinal cord injuries that have impaired lung, arm, and trunk function.

DETAILED DESCRIPTION:
Study Aim 1. This study is aimed to evaluate the effects of non-invasive transcutaneous electrical spinal-cord stimulation (TcESCS) applied below the neurological level of Spinal Cord Injury (SCI) on respiratory, upper extremity, and trunk functional and motor control properties and identify their underlying physiological mechanisms. Evaluation of the mechanisms of respiratory and motor control modulations evoked by the TcESCS will have important implications for the development of specific therapeutic strategies to fight complications of SCI. The objective of Aim 1 is to investigate whether TcESCS can significantly increase activation of motor networks. This work will be done by electrophysiological characterization of respiratory and other motor responses as assessed at rest and in response to the respiratory and other challenges in SCI individuals. Changes in functional measures will be assessed when the TcESCS device is turned "off" and "on". To evaluate "dose-dependent" effects, changes in surface electromyographic (sEMG) magnitude and muscle co-activation will be assessed when stimulation parameters and location are changed during respiratory efforts and motor tasks. The extent to which the stimulation is associated with the largest change in respiratory and sEMG parameters will be implemented as a strategy to be used during stimulation in combination with Respiratory Training (RT), Arm Training (AT), and Trunk Training (TT). To attain the objective of this aim, we will test the working hypothesis that TcESCS excites specific motor networks leading to amplified motor responses. We will test this hypothesis by applying TcESCS during our original approach of the Respiratory Motor Control Assessment (RMCA) and other sEMG-based assessments with kinematics to characterize respiratory, arm, and trunk motor function. During these assessments, beat-to-beat Blood Pressure/ Heart Rate (BP/HR), and respiratory rate will be recorded to evaluate respiratory-cardiovascular responses. The rationale for this aim is that successful completion of the proposed research will contribute fundamental elements to our basic knowledge, without which the therapeutic value of TcESCS cannot be understood. The acquisition of such knowledge is critical to the development of specific rehabilitative strategies. When the proposed studies for Aim 1 have been completed, we expect that motor and inter-related characteristics affected by TcESCS in patients with SCI will be established. Such findings would be important because it will allow us, for the first time, to evaluate the ability of non-invasive spinal cord stimulation to enhance the decreased state of spinal network activity thus demonstrating the potential for rehabilitation.

Study Aim 2. The goal is to evaluate the effectiveness and therapeutic mechanisms of the TcESCS combined with task-specific (Respiratory Training) and non-task-specific (Arm Training and Trunk Training) interventions for breathing. Identification of the physiological effects of potential rehabilitative approaches will have important implications for the development of specific therapeutic strategies. The objective of Aim 2 is to investigate the therapeutic effects of RT regimen in combination with TcESCS. This work will be done by using methods outlined in Aim 1 and additional clinical measures all assessed before training, and repeatedly during follow-up period. Working hypothesis that compare to RT alone and TcESCS alone, RT assisted by TcESCS leads to enhanced use-dependent plasticity of respiratory motor networks, leading the functional recovery will be tested by using the approach of detecting changes in respiratory and other motor control outcome measures in response to stimulation and training. The rationale for this aim is that successful completion of the proposed research will advance the field by providing new avenues for the application of activity-based therapy accompanied by the spinal cord stimulation. When the proposed studies for Aim 2 have been completed, it is expected that the rehabilitative capacity of RT with TcESCS will be determined. Such results are important, because, for the first time, identified therapeutic mechanisms of TcESCS will provide evidence that this intervention can enhance the effects of activity-based therapy in participants with SCI.

ELIGIBILITY:
All SCI research participants, irrespective of gender, will be selected based on the following:

Inclusion Criteria:

1. At least 18 years of age at the time of enrollment;
2. Stable medical condition;
3. Non-progressive SCI T5 or above;
4. Sustained SCI at least 12 months prior to enrollment;
5. At least a 15% deficit in pulmonary function outcomes (FVC or FEV1) as was detected by screening spirometry

Exclusion Criteria:

1. Untreated musculoskeletal dysfunction;
2. Unhealed fracture;
3. Untreated contracture or pressure sore;
4. Ventilator dependence;
5. Untreated depression, psychiatric disorder, or ongoing drug abuse;
6. Major pulmonary or cardiovascular disease;
7. Major esophageal or gastrointestinal disease;
8. Endocrine disorder, malignancy, marked obesity, deep vein thrombosis, or HIV/AIDS related illness;
9. Secondary causes of orthostatic hypotension (anemia, hypervolemia, endocrine, or neurological);
10. Pregnancy by self-report.

All Non-Disabled research participants, irrespective of gender, will be selected based on the following:

Inclusion Criteria:

1. At least 21 years of age at the time of enrollment.
2. FVC and FEV1 values 80% of predicted or above indicating healthy pulmonary function by screening spirometry.

Exclusion Criteria:

1. History of respiratory disease by self-report,
2. History of cardiovascular disease by self-report.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2018-05-17 (Actual); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Non-invasive respiratory electromyography | Through study completion, an average of 1 year.
  Respiratory muscle activity evaluated using vector analysis outcome measure.
Spirometry | Through study completion, an average of 1 year.
  Respiratory activity evaluated using airflow outcome measure.
Maximum airway pressure | Through study completion, an average of 1 year.
  Respiratory activity evaluated using airway pressure measurement.

SECONDARY OUTCOMES:
Functional Neurophysiological Assessment (FNPA) | Through study completion, an average of 1 year.
  The FNPA assesses the motor capacity and control of the upper and lower extremities and trunk .
Multisegmental Motor Response (MMR) | Through study completion, an average of 1 year.
  MMRs in response to non-invasive stimulation of the dorsal spinal cord assessed electromyographically
Transcranial Magnetic Stimulation (TMS) | Through study completion, an average of 1 year.
  TMS of the cortex to assess the integrity of the descending corticospinal tracts
Aerobic Endurance Test (VO2Peak) | Through study completion, an average of 1 year.
  Oxygen consumption during exercise
Spinal Cord Independence Measure (SCIM) | Through study completion, an average of 1 year.
  Questionnaire to assess Self-Care and Mobility
The Craig Handicap Assessment & Reporting Technique (CHART) | Through study completion, an average of 1 year.
  Questionnaire to measure the level of handicap in a community setting: physical independence, mobility, occupation, social integration, and economic self-sufficiency
Beat-by-beat arterial blood pressure | During assessments.
  Non-invasive blood pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Ovechkin, MD, PhD, Principal Investigator — University of Louisville
Locations (1):
- Frazier Rehabilitation and Neuroscience Institute, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gerasimenko Y, Gorodnichev R, Moshonkina T, Sayenko D, Gad P, Reggie Edgerton V. Transcutaneous electrical spinal-cord stimulation in humans. Ann Phys Rehabil Med. 2015 Sep;58(4):225-231. doi: 10.1016/j.rehab.2015.05.003. Epub 2015 Jul 20. PMID 26205686